CLINICAL TRIAL: NCT05314348
Title: Exploring the Electro-mechanical Coupling of Fasciculations in Motor Neuron Disease Using Surface Electromyography and Ultrasound: a Feasibility Study
Brief Title: Surface EMG and Ultrasound in MND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCH19-072
Record Dates: First submitted 2019-08-20; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: 12 MND/ALS patients and 13 healthy controls to be assessed at a single time-point each
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Neuron Disease (Active Comparator): High-density surface EMG Ultrasound
  Interventions: Device: High-density surface EMG; Device: Ultrasound
- Healthy controls (Active Comparator): High-density surface EMG Ultrasound
  Interventions: Device: High-density surface EMG; Device: Ultrasound

INTERVENTIONS:
Device: High-density surface EMG — High-density surface EMG for fasciculation detection
Device: Ultrasound — Ultrasound for fasciculation detection

SUMMARY:
Patients with motor neurone disease typically experience relentless motor decline and die within three years of symptom onset from respiratory muscle weakness. There are currently no effective therapies and the discovery of novel therapies is hampered by the lack of a sensitive disease biomarker. Consequently, there is a huge drive to discover novel biomarkers, which can reliably track disease progression over time. These can then be incorporated into clinical drug trials to expedite effective drug discovery.

Muscle fasciculations represent the hyperexcitability of diseased motor neurons and are almost universally present from the early stages of MND. We predict that the site, frequency and shape of fasciculations might provide a sensitive measure of disease progression in an individual.

We have been conducting a 12-month longitudinal study of 25 patients, performing high-density surface EMG every two months. We have validated an automated technique to process these large data sets. Ultrasound is widely used in clinical medicine to assess anatomical structure in a safe and non-invasive way. Dr Emma Hodson-Tole (Manchester Metropolitan University) and her group have been applying this to the analysis of fasciculations in healthy individuals and patients with MND.

This collaborative project will explore combining these two techniques simultaneously in patients with motor neuron disease and control subjects. The goal is to explore the nature of electro-mechanical coupling related to fasciculations and to determine whether any of these properties are pathophysiological. This would complement other studies from our two groups, investigating the natural history and potential utility of fasciculations as a biomarker of motor neuron health in MND.

ELIGIBILITY:
Inclusion criteria for MND patients:

(i) Aged between 40 and 80 years of age inclusive, at the time of signing the informed consent.

(ii) Diagnosed with MND by a neurologist with expertise in MND. For subjects with bulbar onset there must be objective limb involvement of at least one limb. (iii) Diagnosed with MND within 24 months of symptom onset. (iv) Subjects must be ambulatory (i.e. must not be confined to a wheelchair). (v) Male and female subjects (vi) Capable of giving signed (or verbal consent or assent where applicable) informed consent as described in Protocol Section 9.2 which includes compliance with the requirements and restrictions listed in the consent form and in the protocol. (vii) Capable and willing to comply with the requirements of the protocol (either by themselves or with assistance).

Inclusion criteria for healthy controls (i) Aged between 40 and 80 years of age inclusive, at the time of signing the informed consent.

(ii) Male and female subjects (vi) Capable of giving signed (or verbal consent or assent where applicable) informed consent as described in Protocol Section 9.2 which includes compliance with the requirements and restrictions listed in the consent form and in the protocol. (vii) Capable and willing to comply with the requirements of the protocol

Exclusion criteria for MND patients:

(i) Neurological (other than the subject's MND) or non neurological co morbidities (e.g. joint disease, respiratory disease) which limit mobility.

(ii) Clinically significant cognitive impairment in the opinion of the investigator or lacking capacity in accordance with the Mental Capacity Act (2005).

(iii) Regionally restricted forms of MND, or other atypical variants:

* Isolated corticobulbar pattern of MND with normal ambulation
* Primary lateral sclerosis
* Signs of chronic partial denervation restricted to a single limb
* MND or parkinsonism dementia complex (iv) Subjects requiring mechanical ventilation (non invasive ventilation for sleep apnoea is allowed).

  (v) Historical or current evidence of clinically significant uncontrolled disease which, in the opinion of the chief investigator, would put the safety of the subject at risk through participation or impact the study assessments or endpoints. (vi) Presence of an active implantable cardiac medical device (e.g., pacemaker or implantable cardioverter defibrillator) or at a high risk for needing external defibrillation.

(vii) History of skin hypersensitivity to adhesives. (viii) Current participation in a clinical trial which in the opinion of the chief investigator might impact the objectives of this study.

Exclusion criteria for healthy participants:

(i) Historical or current evidence of clinically significant uncontrolled disease which, in the opinion of the chief investigator, would put the safety of the subject at risk through participation or impact the study assessments or endpoints. (ii) Presence of an active implantable cardiac medical device (e.g., pacemaker or implantable cardioverter defibrillator) or at a high risk for needing external defibrillation.

(iii) History of skin hypersensitivity to adhesives. (iv) Current participation in a clinical trial which in the opinion of the chief investigator might impact the objectives of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between automated detection of fasciculations by two methods (high-density surface EMG and ultrasound) | Single time-point

SECONDARY OUTCOMES:
To assess the practical feasibility of using high-density surface EMG and ultrasound simultaneously in biceps and gastrocnemius. | Single time-point
To highlight potential biomarkers of disease related to the electromechanical coupling of fasciculations (e.g. latency between electrical and mechanical peaks). | Single time-point

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bashford J, Wickham A, Iniesta R, Drakakis E, Boutelle M, Mills K, Shaw C. SPiQE: An automated analytical tool for detecting and characterising fasciculations in amyotrophic lateral sclerosis. Clin Neurophysiol. 2019 Jul;130(7):1083-1090. doi: 10.1016/j.clinph.2019.03.032. Epub 2019 Apr 19. PMID 31078984
- [Background] Bibbings K, Harding PJ, Loram ID, Combes N, Hodson-Tole EF. Foreground Detection Analysis of Ultrasound Image Sequences Identifies Markers of Motor Neurone Disease across Diagnostically Relevant Skeletal Muscles. Ultrasound Med Biol. 2019 May;45(5):1164-1175. doi: 10.1016/j.ultrasmedbio.2019.01.018. Epub 2019 Mar 8. PMID 30857760